CLINICAL TRIAL: NCT06530472
Title: The Relationship Between Belief, Expectation, and Adherence to Therapy During COVID-19 Pandemic: a Multigroup Cohort Study in Patients With Ischemic Heart Disease
Brief Title: The Relationship Between Belief, Expectation, and Adherence to Therapy During COVID-19 Pandemic
Acronym: RACAT-COVID
Status: Enrolling by invitation | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Ospedale Valduce, Como (Unknown); Azienda Ospedaliera Niguarda Cà Granda (Other)
Responsible Party: Sponsor
Other Study IDs: FDG_88-15
Record Dates: First submitted 2024-07-29; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-02

CONDITIONS: Ischemic Heart Diseases
Keywords: Ischemic Heart Disease; Adherence; Belief; Acceptance; COVID-19
MeSH Terms: conditions — Myocardial Ischemia; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fondazione Don Carlo Gnocchi: All patients diagnosed with ischaemic heart disease established by angiography; attained age of majority; Score >= 26 on the Montreal Cognitive Assessment (MoCA) test. At baseline, 3, 6 and 12 months, people will undergo to both a psychological and cardiological assessment.
  Interventions: Other: Monitoring
- Ospedale Valduce: All patients diagnosed with ischaemic heart disease established by angiography; attained age of majority; Score >= 26 on the Montreal Cognitive Assessment (MoCA) test. At baseline, 3, 6 and 12 months, people will undergo to both a psychological and cardiological assessment.
  Interventions: Other: Monitoring
- Ospedale Cà Granda Niguarda: All patients diagnosed with ischaemic heart disease established by angiography; attained age of majority; Score >= 26 on the Montreal Cognitive Assessment (MoCA) test. At baseline, 3, 6 and 12 months, people will undergo to both a psychological and cardiological assessment.
  Interventions: Other: Monitoring

INTERVENTIONS:
Other: Monitoring — At baseline, 3, 6 and 12 months, people will undergo to both a psychological and cardiological assessment.

SUMMARY:
The goal of this [type of study: observational study or clinical trial ] is to learn about, test, compare etc.] in [ describe participant population/health conditions ]. The main question [ it aims to answer are:

* [question
* [question Participants will [describe the main tasks participants will be asked to do, treatments they'll be given and use bullets if it is more than 2 items ].

If there is a comparison group: Researchers will compare insert groups ] to see if insert effects

ELIGIBILITY:
Inclusion Criteria:

* all patients diagnosed with ischaemic heart disease established by angiography;
* reaching the age of majority;
* score >= 26 on the Montreal Cognitive Assessment (MoCA) test (Nasreddine et al., 2005).

Exclusion Criteria:

* presence of comorbidity with other pathologies in an active or advanced phase; -patients with a prognosis to be defined;
* pregnancy;
* participants with neurological pathologies that significantly impair their cognitive functions (e.g. advanced Parkinson's disease; Alzheimer's dementia...cardiac arrest with hypoxic damage);
* participants with cognitive impairments that compromise comprehension and sharing of the contents of the questions, detected through the administration of the Montreal Cognitive Assessment (MoCA) test (Nasreddine et al., 2005).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with ischaemic heart disease established by angiography
Sampling Method: Non-Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Adherence | At baseline, 3, 6 and 12 months from the recruitment
  Measured by the percentage of days covered (Percentage of Days Covered, PDC) by antiplatelet therapy, beta-blockers, statins, ACE-I/Sartan, hypoglycaemic drugs, psychotropic drugs (anxiolytics; antidepressants).
  The PDC is defined as the proportion of days for which a patient has a supply of medication available. When multiple prescriptions are for the same day, reference is made to the maximum duration, and for overlapping prescriptions, sequential use of the two prescriptions is assumed by summing the days of supply for each. Any interruptions in therapy are also taken into account. Non-adherence is defined as a PDC of less than 80%, while non-persistence is defined as a gap in prescriptions of (Direct Oral Anticoagulants or Direct Oral Anticoagulants) DOACs ≥14 days (Yu et al., 2020).
NACE | At baseline, 3, 6 and 12 months from the recruitment
  Net adverse clinical event or NACE, defined as a composite of all-cause mortality, myocardial infarction, stroke or major haemorrhage. In this case, bleeding is definitive according to the BARC (Bleeding Academic Research Consortium) scale (Mehran et al., 2011).
MARS-i | At baseline, 3, 6 and 12 months from the recruitment
  Measure with theMARS-5-i questionnaire consists of five questions on forgetting, changing dosage, stopping, skipping, and taking less medication . The score ranges from 5 to 25, where a higher MARS-5-i score indicates higher self-reported adherence. One item assesses unintentional non-adherence and four items assess intentional non-adherence

SECONDARY OUTCOMES:
Extra visits | At baseline, 3, 6 and 12 months from the recruitment
  Number of extra (unplanned) visits, frequency of planned follow-up visits
Adherence to pharmacotherapy | At baseline, 3, 6 and 12 months from the recruitment
  Measured as difference between number of pills taken and number of pills prescribed.
  At each time of data collection, monitoring will be carried out for all four recommended therapies in patients with reduced ejection fraction (entero, jardiance, beta blockade, anti-aldosterone).
  It is also intended to detect how many patients, at one year, have optimal control of risk factors, in terms of lipid profile at target, glycaemic control, smoking cessation, maintenance of regular physical activity, BMI improvement (considering LDL value, fasting blood glucose, HbA1 for diabetics).
CAS | At baseline, 3, 6 and 12 months from the recruitment
  Measured by the Coronavirus Anxiety Scale (CAS) (Lee, 2020; Silva et al., 2020), which assesses dysfunctional anxiety associated with the Covid-19 crisis. Each item on the CAS is rated on a 5-point scale, from 0 (not at all) to 4 (almost every day), based on experiences over the past two weeks. This scale format is consistent with the DSM-5 measure of cross-sectional symptoms. A total CAS score ≥ 9 indicates probable coronavirus-related dysfunctional anxiety. High scores on a particular item or a high total scale score (≥ 9) may indicate problematic symptoms for the individual that may warrant further assessment and/or treatment. Clinical judgement should guide the interpretation of CAS results.
CSS | At baseline, 3, 6 and 12 months from the recruitment
  Measured by the Covid-19 Stress Scale (CSS) (Taylor et al., 2020), a 36-item scale developed to better understand and assess Covid-19-related distress. The subscales assess symptoms of Covid-related stress and anxiety: (1) fear of danger and contamination, (2) fear of economic consequences, (3) xenophobia, (4) compulsive control and reassurance seeking, and (5) symptoms of traumatic stress on Covid-19. The scales were found to be robust on various reliability and validity indices. The scales are intercorrelated, providing evidence of a Covid-19-related stress syndrome. The scales are promising as tools to better understand the distress associated with Covid-19 and to identify persons in need of mental health services.
BIPQ | At baseline, 3, 6 and 12 months from the recruitment
  Detected with the Brief Illness Perception Questionnaire (BIPQ) (Broadbent et al., 2006), a nine-item scale designed to rapidly assess cognitive and emotional representations of illness.
ICQ | At baseline, 3, 6 and 12 months from the recruitment
  Illness Cognition Questionnaire (ICQ) (Evers et al., 2001), which evaluates three ways of cognitively assessing the stressful and adverse nature of a chronic illness: helplessness, acceptance and perceived benefits.
Anxiety | At baseline, 3, 6 and 12 months from the recruitment
  Measured through the use of the Hospital Anxiety and Depression Scale (HADS) test (Zigmond & Snaith, 1983), a widely used instrument to measure psychological morbidity in chronically ill patients, which consists of 14 items designed to detect the presence of anxiety and depression.
Depression | At baseline, 3, 6 and 12 months from the recruitment
  Measured through the use of the Hospital Anxiety and Depression Scale (HADS) test (Zigmond & Snaith, 1983), a widely used instrument to measure psychological morbidity in chronically ill patients, which consists of 14 items designed to detect the presence of anxiety and depression.
Illness Expectations | At baseline, 3, 6 and 12 months from the recruitment
  Some questions specifically formulated to assess explicit disease expectations in heart disease are proposed. These questions will be integrated by the administration of a semi-structured interview.
Socio-demographic data | At baseline
  Date of birth, gender, education, current or previous occupation, marital status, presence of children, smoking, physical activity, presence of heart disease in the family.
Clinical data | At baseline, 3, 6 and 12 months from the recruitment
  Weight and height (for the calculation of Body Mass Index, BMI), blood pressure, heart rate, oxygen saturation, blood test results (complete lipid profile, blood glucose, glycated haemoglobin), co-morbidities, perceived symptoms (breathlessness, chest pressure, angina pectoris, sweating, fainting, nausea, vomiting) acute or elective indication for surgery (specify if patient treated percutaneously or cardiac surgery); post-acute destination (patient discharged home, started on a rehabilitation programme, other); haemodialysis; PCSK9; left ventricular ejection fraction data; reports (coronary angiography, echocardiogram), having contracted Covid-19; presence of asthenia and/or dyspnoea.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Evers AW, Kraaimaat FW, van Lankveld W, Jongen PJ, Jacobs JW, Bijlsma JW. Beyond unfavorable thinking: the illness cognition questionnaire for chronic diseases. J Consult Clin Psychol. 2001 Dec;69(6):1026-36. PMID 11777106
- [Background] Miyazaki M, Nakashima A, Nakamura Y, Sakamoto Y, Matsuo K, Goto M, Uchiyama M, Okamura K, Mitsutake R, Urata H, Kamimura H, Imakyure O. Association between medication adherence and illness perceptions in atrial fibrillation patients treated with direct oral anticoagulants: An observational cross-sectional pilot study. PLoS One. 2018 Sep 28;13(9):e0204814. doi: 10.1371/journal.pone.0204814. eCollection 2018. PMID 30265710
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372